CLINICAL TRIAL: NCT05220475
Title: A Comparison of a Fully Covered Self-expandable Metal Stent With an External Anchoring Plastic Stent and Uncovered Stent: Prospective Randomized Multicenter Study
Brief Title: A Comparison of a Fully Covered Self-expandable Metal Stent With an External Anchoring Plastic Stent and Uncovered Stent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Hyub Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2012-043-1179
Record Dates: First submitted 2022-01-04; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Malignant Biliary Obstruction
Keywords: Fully Covered Self Expandable Metal Stent; Uncovered Self Expandable Metal Stent

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- fc-SEMS with anchoring plastic stent (Experimental): fully covered self-expanable metal stent with an external anchoring plastic stent
  Interventions: Device: fully covered self-expandable metal stent with an anchoring external plastic stent
- uc-SEMS (Active Comparator): uncovered self-expandable metal stent
  Interventions: Device: uncovered self-expandable metal stent

INTERVENTIONS:
Device: fully covered self-expandable metal stent with an anchoring external plastic stent — Extrahepatic malignant biliary obstruction treated with fully covered self-expandable metal stent with an anchoring plastic stent
  Arms: fc-SEMS with anchoring plastic stent
Device: uncovered self-expandable metal stent — Extrahepatic malignant biliary obstruction treated with uncovered self-expandable metal stent without an anchoring plastic stent
  Arms: uc-SEMS

SUMMARY:
Multi-center, randomized controlled study fc-SEMS with anchoring plastic stent vs uc-SEMS in malignant biliary obstruction

DETAILED DESCRIPTION:
This study is multi-center, randomized controlled study to compare the stent patency in malignant biliary obstruction. The patency of fully covered self expandable metal stent with external anchoring plastic stent was compared with that of uncovered self expandable metal stent.

ELIGIBILITY:
Inclusion Criteria:

* Adults with 19 years of age or older
* Those who voluntarily consented to the trial and signed a written consent
* Inoperable malignant biliary obstruction

Exclusion Criteria:

* Previous surgical biliary drainage
* Patients continuosly requiring percutaneous transhepatic biliary drainage
* History of biliary drainage with metal stent
* Biliary obstruction located in hilum or intrahepatic duct
* Patients with life expectancy of 3 months or less
* On pregnancy
* Unable to underwent endoscopic procedures

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-10-24 (Estimated); Study Completion 2024-10-24 (Estimated)

PRIMARY OUTCOMES:
Rate of patent stent | 1 year
  The number of patient without stent dysfuction divided by total number of patients

SECONDARY OUTCOMES:
Stent obstruction | 1 year
  Suspected by jaundice (Total bilirubin > 2 upper normal limit) or radiologic finding of stent occlusion which is confirmed by ERCP
Stent migration | 1 year
  Radiologic finding of migration through Abdomen X-ray or CT scan
Re-intervention | 1 year
  Endoscopic retrograde biliary drainage or Percutaneous transhepatic biliary drainage
Adverse event | 1 year
  acute cholangitis, acute cholecystitis, acute pancreatitis
Overall survival | 1 year
  Timespan from the diagnosis to the death

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hyub Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea